CLINICAL TRIAL: NCT07239427
Title: Use of Transcranial Direct Current Stimulation (TDCS) in an Active Pain Coping Program for Patients With Fibromyalgia: A Randomized Control Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Manuel Santos Bermejo, MSc, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI-25-574-APE
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Transcranial Direct Current Stimulation; Neuromodulation; Therapeutic Exercise; Pain Science Education; Pain Neuroscience Education
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are masked (blinded): Participants are unaware of their group assignment, as the control group receives a sham Transcranial Direct Current Stimulation (tDCS) protocol that is designed to be indistinguishable from the active stimulation.
  Investigators are masked (blinded): The study personnel responsible for collecting the primary outcome data and performing the statistical analysis will also be masked (blinded) to the participants' group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS and Multimodal Active Pain Coping Program (Experimental): This group receives the Multimodal Active Pain Coping Program. The intervention sequence is: 8 sessions of Pain Neuroscience Education (PNE), followed by 5 daily sessions of Active Transcranial Direct Current Stimulation (tDCS), and then 18 sessions of Therapeutic Exercise (TE). The Active tDCS is applied over the primary motor cortex (M1) and orbitofrontal region for 20 minutes at 2 mA, aiming to potentiate the analgesic effects of the overall Active Pain Coping strategies.
  Interventions: Behavioral: Pain Science Education; Device: Transcranial Direct Current Stimulation; Behavioral: Therapeutic Exercise
- Sham tDCS and Multimodal Active Pain Coping Program (Sham Comparator): This group receives the identical Multimodal Active Pain Coping Program. The intervention sequence is: 8 sessions of Pain Neuroscience Education (PNE), followed by 5 daily sessions of Sham (Placebo) Transcranial Direct Current Stimulation (tDCS), and then 18 sessions of Therapeutic Exercise (TE). The Sham tDCS uses the same electrode placement but only runs for a few seconds to maintain participant blinding, providing no active current for the remainder of the 20-minute session.
  Interventions: Behavioral: Pain Science Education; Behavioral: Therapeutic Exercise; Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Behavioral: Pain Science Education — Pain Science Education component is the initial phase of the multimodal Active Pain Coping program. Its objective is to reframe maladaptive beliefs about pain in Fibromyalgia patients by providing a modern neuroscientific understanding of their persistent pain condition. The content focuses on explaining that pain does not necessarily equate to tissue damage but is a protective output generated by the brain, addressing the physiology of pain and sensitization, the relationship between fear and movement avoidance (kinesiophobia), and the potential of neuroplasticity to "retrain" the nervous system. This phase is crucial for reducing pain catastrophizing and fear, thereby empowering the patient to actively and fully participate in the subsequent treatment phases.
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) is a non-invasive neuromodulation technique used in this study to enhance the central analgesic effects of the combined Active Pain Coping treatment. The intervention involves the delivery of a low-intensity electrical current through the scalp to modulate cortical excitability. The Anode is positioned over the Primary Motor Cortex (M1) (C3) and the Cathode is placed over the Orbitofrontal region (FP2). The Active Group receives a constant 2 mA current for 20 minutes to modulate brain activity.
  Arms: Active tDCS and Multimodal Active Pain Coping Program
Behavioral: Therapeutic Exercise — Therapeutic Exercise (TE) is the most extensive component of the multimodal program, administered in structured group sessions lasting approximately one hour. The protocol is designed to be adapted to each patient's physical condition, and includes a graded exposure component to ensure safety and mitigate pain flares. Each session includes a warm-up (mobility/activation); a main phase focused on conscious movement, coordination, balance, agility, and muscular strength; and a final cool-down that incorporates flexibility, relaxation, and mindfulness. The primary purpose of this structured exercise is to safely promote physical activity, reverse physical deconditioning and muscle atrophy, reduce fear of movement (kinesiophobia), and reinforce the new neuroscientific understanding of pain acquired, thereby sustaining the overall analgesic effects of the treatment.
Device: Sham Transcranial Direct Current Stimulation — Control Group receives an identical-looking Sham (Placebo) stimulation, where the device runs for only the initial minute (at 2 mA) before turning off silently, ensuring the participants remain blinded to the treatment they receive.
  Arms: Sham tDCS and Multimodal Active Pain Coping Program

SUMMARY:
The trial is designed to determine the added effect of active transcranial direct current stimulation (tDCS) when combined with a multimodal Active Pain Coping Program in individuals with fibromyalgia. The primary objective is to compare the effectiveness of active versus sham tDCS when both are delivered to the same standardized multimodal intervention. All participants will undergo an identical treatment sequence consisting of 8 sessions of Pain Neuroscience Education (PNE), followed by 5 consecutive daily sessions of either active or sham tDCS, and 18 sessions of therapeutic exercise (TE). Active tDCS will be administered over the primary motor cortex (M1) and orbitofrontal region for 20 minutes at 2 mA. The sham procedure will replicate the electrode placement and brief initial stimulation to ensure blinding, with no active current thereafter. Secondary outcomes will examine changes in pain intensity, central pain processing, psychological variables, and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Must have a prior diagnosis of Fibromyalgia (FM), which must be documented and validated in the patient's medical record.

Exclusion Criteria:

* Neurological Conditions: History of epilepsy or any other decompensated neurological condition that could contraindicate Transcranial Direct Current Stimulation (tDCS).
* Active Pathologies: Presence of other active or recent pathologies (e.g., cancer, fractures, fissures, or severe traumatic accidents of the skull) that could interfere with treatment or evaluation.
* Pregnancy: Currently pregnant or planning to become pregnant during the study period.
* Metallic Implants: Presence of metallic implants in the skull that may interact with or contraindicate the use of tDCS.
* Concurrent Studies: Active participation in another concurrent clinical research study involving treatments for fibromyalgia.
* Protocol Adherence: Inability to understand or adhere to the treatment and evaluation protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Outcome measures will be assessed at baseline (enrollment), post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  The Fibromyalgia Impact Questionnaire (FIQ) assesses the global impact and severity of FM across 10 items covering Physical Function, Work Status, and Symptoms (pain, fatigue, stiffness, etc.). The total score ranges from 0 to 100.
  The calculation involves summing and scaling the scores from the three components: Physical Function is scored on a 4-point scale (0-3) and the sum is then multiplied by 3; Work Status and Symptoms (rated on VAS/NRS) are scaled to contribute to the final 100-point total.
  The FIQ is a disability and severity index: a higher score (closer to 100) indicates a greater impact of fibromyalgia, signifying higher functional disability, more severe symptoms, and a worse quality of life. Conversely, a lower score (closer to 0) indicates a better health status. The primary objective is to observe a significant decrease in this score.

SECONDARY OUTCOMES:
Pain Intensity (Visual analogue scale) | Baseline, Post-Intervention (12 weeks), and Follow-up (6 months).
  Measures the current subjective pain level reported by the patient. Score of the Visual/Numeric Analog Scale (0 to 10).
Conditioned Pain Modulation (CPM) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  The Conditioned Pain Modulation (CPM) test is used to assess the central nervous system's capacity for endogenous pain inhibition. Using a parallel paradigm, a Test Stimulus (T-Test), which measures the baseline Pressure Pain Threshold (PPT), is measured simultaneously with a Conditioning Stimulus (C-Test). The C-Test is applied by inflating a blood pressure cuff to induce ischemia in the contralateral limb. The pain threshold is then measured again at the T-Test site while the ischemic stimulus is active. The CPM effect is quantified as the change (either the absolute difference or percentage change) in the PPT measured during the ischemic stimulation compared to the baseline PPT, where an increase in the threshold indicates effective CPM.
Pressure Pain Thresholds (PPT) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  Pressure Pain Thresholds (PPTs) are measured using a Wagner brand Fisher digital algometer to quantify local pain sensitivity in $\text{kg/cm}^2$. Measurements are taken at four specific anatomical reference points bilaterally: the midpoint between the posterior border of the acromion and the C7 spinal process, and the midpoint between the highest part of the superior border of the iliac crest and the spinal process at the same height. At each point, two consecutive measurements are taken by increasing pressure at a rate of $1\text{ kg/cm}^2$ per second. The threshold is determined when the participant reports that the sensation of pressure turns into pain. The final PPT score for each site is the average of the two consecutive measurements. A lower PPT indicates increased local pain sensitivity.
Change in Temporal Summation | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  Temporal Summation (TS) is used to assess central sensitization (the wind-up phenomenon). It is provoked by applying 10 consecutive pulses using a pressure algometer at the previously determined Pressure Pain Threshold (PPT) for the specific location. For each pulse, pressure is gradually increased at a rate of 2kg/s to reach the PPT, held for 1 second, and then released with a 1-second interval before the next pulse. The participant rates the pain intensity of the first, fifth, and tenth pulse on a Numerical Rating Scale (NRS) from 0 (no pain) to 10 (worst possible pain). A score increase between the first and tenth pulse indicates efficient temporal summation (central sensitization).
Pain Catastrophizing Scale (PCS) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  The Pain Catastrophizing Scale (PCS) is a 13-item psychometric tool used to assess negative cognitive and emotional responses related to actual or anticipated pain. The scale evaluates three subcomponents: Rumination (inability to stop focusing on pain), Magnification (exaggerating the threat of pain), and Helplessness (feeling unable to cope with the pain).
  Each of the 13 items is rated on a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("all the time").
  The total score is calculated by summing the scores from all 13 items, resulting in a final score that ranges from 0 to 52. A higher score on the PCS indicates greater pain catastrophizing (a worse cognitive outcome), which is strongly associated with increased pain intensity and functional disability.
Hospital Anxiety and Depression Scale (HADS) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item screening tool used to assess the severity of Anxiety and Depression symptoms in medical patients, avoiding confounding physical symptoms. It comprises two subscales: HADS-A (Anxiety) and HADS-D (Depression), each containing 7 intermingled items. Each item is rated on a 4-point Likert scale ranging from 0 ("not at all") to 3 ("most of the time"). The total score for each separate subscale ranges from 0 to 21. A higher score on either the HADS-A or HADS-D subscale indicates greater severity of anxiety or depressive symptoms, respectively. Scores are used both as continuous variables and often categorized for clinical interpretation.
Tampa Scale Kinesiophobia (TSK-11) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  The Tampa Scale for Kinesiophobia (TSK-11) is an 11-item tool used to assess fear of movement, injury, or re-injury (kinesiophobia). It specifically evaluates the patient's belief that physical activity is dangerous or harmful. Each of the 11 items is scored on a 4-point Likert scale, ranging from 1 ("strongly disagree") to 4 ("strongly agree"). The total score is calculated by summing the scores from all 11 items, with some items being reverse-scored to maintain consistency. The final score ranges from 11 to 44. A higher total score on the TSK-11 indicates greater kinesiophobia and subsequent avoidance behaviors, which are linked to increased pain intensity and functional disability in chronic pain populations.
Medical Outcomes Study Sleep Scale (MOS SS) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  12-item questionnaire that assesses a person's sleep quality and problems over a four-week period. It measures six key areas: sleep disturbance, sleep adequacy, somnolence (daytime sleepiness), snoring, waking due to shortness of breath or headache, and quantity of sleep. The scale yields scores for these six domains, as well as two global sleep problem indices
International Physical Activity Questionnaire (IPAQ) | Baseline, post-intervention (end of the 12-week treatment protocol), and at a 3-month follow-up after treatment.
  The International Physical Activity Questionnaire (IPAQ) is a standardized tool that defines and measures physical activity based on frequency and duration over a week. It categorizes physical activity into vigorous-intensity, moderate-intensity, and walking, and also assesses time spent sitting. The IPAQ covers activity across different domains, including work, transportation, domestic chores, and leisure time, to provide a comprehensive picture of a person's physical activit

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Estrategias de Afrontamiento Activo del Dolor., Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Staud R, Weyl EE, Riley JL 3rd, Fillingim RB. Slow temporal summation of pain for assessment of central pain sensitivity and clinical pain of fibromyalgia patients. PLoS One. 2014 Feb 18;9(2):e89086. doi: 10.1371/journal.pone.0089086. eCollection 2014. PMID 24558475
- [Result] Staud R, Vierck CJ, Cannon RL, Mauderli AP, Price DD. Abnormal sensitization and temporal summation of second pain (wind-up) in patients with fibromyalgia syndrome. Pain. 2001 Mar;91(1-2):165-75. doi: 10.1016/s0304-3959(00)00432-2. PMID 11240089
- [Result] Sosa-Reina MD, Nunez-Nagy S, Gallego-Izquierdo T, Pecos-Martin D, Monserrat J, Alvarez-Mon M. Effectiveness of Therapeutic Exercise in Fibromyalgia Syndrome: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Biomed Res Int. 2017;2017:2356346. doi: 10.1155/2017/2356346. Epub 2017 Sep 20. PMID 29291206
- [Result] Serrat M, Almirall M, Muste M, Sanabria-Mazo JP, Feliu-Soler A, Mendez-Ulrich JL, Luciano JV, Sanz A. Effectiveness of a Multicomponent Treatment for Fibromyalgia Based on Pain Neuroscience Education, Exercise Therapy, Psychological Support, and Nature Exposure (NAT-FM): A Pragmatic Randomized Controlled Trial. J Clin Med. 2020 Oct 18;9(10):3348. doi: 10.3390/jcm9103348. PMID 33081069
- [Result] Schmidt-Wilcke T, Luerding R, Weigand T, Jurgens T, Schuierer G, Leinisch E, Bogdahn U. Striatal grey matter increase in patients suffering from fibromyalgia--a voxel-based morphometry study. Pain. 2007 Nov;132 Suppl 1:S109-S116. doi: 10.1016/j.pain.2007.05.010. Epub 2007 Jun 22. PMID 17587497
- [Result] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295
- [Result] O'Brien AT, Deitos A, Trinanes Pego Y, Fregni F, Carrillo-de-la-Pena MT. Defective Endogenous Pain Modulation in Fibromyalgia: A Meta-Analysis of Temporal Summation and Conditioned Pain Modulation Paradigms. J Pain. 2018 Aug;19(8):819-836. doi: 10.1016/j.jpain.2018.01.010. Epub 2018 Feb 15. PMID 29454976
- [Result] Mhalla A, de Andrade DC, Baudic S, Perrot S, Bouhassira D. Alteration of cortical excitability in patients with fibromyalgia. Pain. 2010 Jun;149(3):495-500. doi: 10.1016/j.pain.2010.03.009. Epub 2010 Mar 31. PMID 20356675
- [Result] Mhalla A, Baudic S, de Andrade DC, Gautron M, Perrot S, Teixeira MJ, Attal N, Bouhassira D. Long-term maintenance of the analgesic effects of transcranial magnetic stimulation in fibromyalgia. Pain. 2011 Jul;152(7):1478-1485. doi: 10.1016/j.pain.2011.01.034. Epub 2011 Mar 11. PMID 21397400
- [Result] Mendonca ME, Simis M, Grecco LC, Battistella LR, Baptista AF, Fregni F. Transcranial Direct Current Stimulation Combined with Aerobic Exercise to Optimize Analgesic Responses in Fibromyalgia: A Randomized Placebo-Controlled Clinical Trial. Front Hum Neurosci. 2016 Mar 10;10:68. doi: 10.3389/fnhum.2016.00068. eCollection 2016. PMID 27014012
- [Result] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Result] Lutz J, Jager L, de Quervain D, Krauseneck T, Padberg F, Wichnalek M, Beyer A, Stahl R, Zirngibl B, Morhard D, Reiser M, Schelling G. White and gray matter abnormalities in the brain of patients with fibromyalgia: a diffusion-tensor and volumetric imaging study. Arthritis Rheum. 2008 Dec;58(12):3960-9. doi: 10.1002/art.24070. PMID 19035484
- [Result] Lloyd DM, Wittkopf PG, Arendsen LJ, Jones AKP. Is Transcranial Direct Current Stimulation (tDCS) Effective for the Treatment of Pain in Fibromyalgia? A Systematic Review and Meta-Analysis. J Pain. 2020 Nov-Dec;21(11-12):1085-1100. doi: 10.1016/j.jpain.2020.01.003. Epub 2020 Jan 23. PMID 31982685
- [Result] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Result] Knijnik LM, Dussan-Sarria JA, Rozisky JR, Torres IL, Brunoni AR, Fregni F, Caumo W. Repetitive Transcranial Magnetic Stimulation for Fibromyalgia: Systematic Review and Meta-Analysis. Pain Pract. 2016 Mar;16(3):294-304. doi: 10.1111/papr.12276. Epub 2015 Jan 12. PMID 25581213
- [Result] Jensen KB, Loitoile R, Kosek E, Petzke F, Carville S, Fransson P, Marcus H, Williams SC, Choy E, Mainguy Y, Vitton O, Gracely RH, Gollub R, Ingvar M, Kong J. Patients with fibromyalgia display less functional connectivity in the brain's pain inhibitory network. Mol Pain. 2012 Apr 26;8:32. doi: 10.1186/1744-8069-8-32. PMID 22537768
- [Result] Hauser W, Ablin J, Perrot S, Fitzcharles MA. Management of fibromyalgia: practical guides from recent evidence-based guidelines. Pol Arch Intern Med. 2017 Jan 4;127(1):47-56. doi: 10.20452/pamw.3877. Epub 2017 Jan 4. PMID 28075425
- [Result] Garcia-Rios MC, Navarro-Ledesma S, Tapia-Haro RM, Toledano-Moreno S, Casas-Barragan A, Correa-Rodriguez M, Aguilar-Ferrandiz ME. Effectiveness of health education in patients with fibromyalgia: a systematic review. Eur J Phys Rehabil Med. 2019 Apr;55(2):301-313. doi: 10.23736/S1973-9087.19.05524-2. Epub 2019 Jan 28. PMID 30698402
- [Result] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Result] Galan-Martin MA, Montero-Cuadrado F, Lluch-Girbes E, Coca-Lopez MC, Mayo-Iscar A, Cuesta-Vargas A. Pain Neuroscience Education and Physical Therapeutic Exercise for Patients with Chronic Spinal Pain in Spanish Physiotherapy Primary Care: A Pragmatic Randomized Controlled Trial. J Clin Med. 2020 Apr 22;9(4):1201. doi: 10.3390/jcm9041201. PMID 32331323
- [Result] Fertonani A, Miniussi C. Transcranial Electrical Stimulation: What We Know and Do Not Know About Mechanisms. Neuroscientist. 2017 Apr;23(2):109-123. doi: 10.1177/1073858416631966. Epub 2016 Jul 8. PMID 26873962
- [Result] Duarte D, Castelo-Branco LEC, Uygur Kucukseymen E, Fregni F. Developing an optimized strategy with transcranial direct current stimulation to enhance the endogenous pain control system in fibromyalgia. Expert Rev Med Devices. 2018 Dec;15(12):863-873. doi: 10.1080/17434440.2018.1551129. Epub 2018 Dec 3. PMID 30501532
- [Result] Desmeules JA, Cedraschi C, Rapiti E, Baumgartner E, Finckh A, Cohen P, Dayer P, Vischer TL. Neurophysiologic evidence for a central sensitization in patients with fibromyalgia. Arthritis Rheum. 2003 May;48(5):1420-9. doi: 10.1002/art.10893. PMID 12746916
- [Result] Castelo-Branco L, Uygur Kucukseymen E, Duarte D, El-Hagrassy MM, Bonin Pinto C, Gunduz ME, Cardenas-Rojas A, Pacheco-Barrios K, Yang Y, Gonzalez-Mego P, Estudillo-Guerra A, Candido-Santos L, Mesia-Toledo I, Rafferty H, Caumo W, Fregni F. Optimised transcranial direct current stimulation (tDCS) for fibromyalgia-targeting the endogenous pain control system: a randomised, double-blind, factorial clinical trial protocol. BMJ Open. 2019 Oct 30;9(10):e032710. doi: 10.1136/bmjopen-2019-032710. PMID 31672712
- [Result] Cabo-Meseguer A, Cerda-Olmedo G, Trillo-Mata JL. Fibromyalgia: Prevalence, epidemiologic profiles and economic costs. Med Clin (Barc). 2017 Nov 22;149(10):441-448. doi: 10.1016/j.medcli.2017.06.008. Epub 2017 Jul 19. English, Spanish. PMID 28734619